CLINICAL TRIAL: NCT04168983
Title: Study of the Impact of Sophrology on the Pain Felt During a Bone Marrow Aspiration and Biopsy
Brief Title: Impact of Sophrology on the Pain Felt During a Bone Marrow Aspiration and Biopsy
Acronym: BOM-ZEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-A00796-51
Record Dates: First submitted 2019-10-03; First posted 2019-11-19 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Hematologic Diseases; Diagnoses Disease; Pain
MeSH Terms: conditions — Hematologic Diseases; Pain

STUDY DESIGN:
Intervention Model Description: Single centre, comparative, controlled randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care: local anesthesia + nitrous oxide and oxygen administration
- Experimental (Experimental): Usual care: local anesthesia + nitrous oxide and oxygen administration
  In this arm : sophrology is added
  Interventions: Other: sophrology

INTERVENTIONS:
Other: sophrology — Sophrology session provided by a nurse sophrologist in addition to the usual care during BMAB
  Arms: Experimental

SUMMARY:
The bone marrow aspiration and biopsy (BMAB) is an essential and indispensable examination for the diagnosis and the follow-up of the hematological diseases but which remains painful and dread by the patients. Until then it was performed manually using a trocar. It is now practiced most often using a tool (like a small drill), device that pierces through the external iliac bone to extract a bone cylinder that will be analyzed

If the gesture is faster than with the manual method, it remains overall painful and the noise generated by the drill that passes through the periosteum of the iliac bone is impressive for the patient.

Prevention measures to limit pain and anxiety are put in place during the examination: local anesthesia, with or without a lidocaine patch, as well as inhalation of a mixture of nitrous oxide and oxygen (MEOPA®). These, recommended by the "Standards, Options, Recommendation" (SOR) often remain insufficient and are not devoid of undesirable effects.

Despite these precautions, several studies show that the action remains painful and anxiety-provoking.

An exploratory survey carried out in the hematology department of the François Baclesse Center in 2013 confirms these results and specifies that the pain remains present for another 30 minutes after the examination.

The investigators believe that associating a psycho-corporeal technique, as is sophrology, with the usual care, could contribute to the decrease of the threshold of pain and anxiety during the BMAB and avoid the use of a premedication.

The effectiveness of sophrology as a complementary technique in the field of pain prevention in invasive procedures is recognized by observations and clinical results. This complementary therapy, among others, has its place in the hospital.

To date, to investigator's knowledge, there is no published, randomized study evaluating the effectiveness of sophrology on pain in invasive procedures.

The investigators propose a study whose main objective is to evaluate the effectiveness of a session of sophrology on the pain felt during the realization of the BMAB, in patients with hematological malignancy. This session will be provided by a sophrologist nurse This study should include 90 patients undergoing a BMAB over a 24-month period.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old who has been informed of the study and has signed the consent form of the study
* Patient with a malignant hemopathy requiring a BMAB as part of a diagnostic assessment
* Patient who has never had a BMAB before
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patient requiring oral premedication
* Patient with contraindications or intolerance to MEOPA®
* Patient with a history of allergy to local anesthetics
* Patient not understanding French
* Patient with deafness
* Patient with severe cognitive impairment
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) score of the pain felt by the patient during the gesture of performing the BMAB | Baseline
  This is a self-assessment. This scale has two sides. On one side, the patient identifies his pain with a ruler, left (no pain) right (the strongest pain he has ever felt).
  On the other hand, the caregiver raises the corresponding score from 0 to 10. Pain will bemeasured a posteriori (not possible to evaluate during the sophrology sesssion)

SECONDARY OUTCOMES:
Numerical score (NS) of anxiety of the patient before the BMAB | Baseline
  The same scale is used to measure anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Touchet, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No